CLINICAL TRIAL: NCT00064233
Title: A Phase I Dose-Escalation Study To Determine The Safety, Pharmacokinetics, And Pharmacodynamics Of BMS-354825 In The Treatment Of Patients With Chronic Phase Chronic Myelogenous Leukemia Who Have Hematologic Resistance To Imatinib Mesylate (Gleevec
Brief Title: BMS-354825 in Treating Patients With Chronic Phase Chronic Myelogenous Leukemia That Is Resistant to Imatinib Mesylate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000310142; UCLA-0303035; BMS-CA180002
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-08

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: dasatinib

SUMMARY:
RATIONALE: BMS-354825 may stop the growth of cancer cells by stopping the enzymes necessary for cancer cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of BMS-354825 in treating patients with chronic phase chronic myelogenous leukemia that is resistant to imatinib mesylate.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose, maximum administered dose, dose-limiting toxicity, and a recommended phase II dose of BMS-354825 in patients with chronic phase chronic myelogenous leukemia who have hematologic resistance to imatinib mesylate.
* Determine the safety and tolerability of this drug in these patients.
* Determine the plasma pharmacokinetics of this drug in these patients.
* Determine, preliminarily, the efficacy of this drug, in terms of hematologic, cytogenetic, and molecular responses in these patients.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive oral BMS-354825 once daily on days 1-5. Courses repeat every 7 days for at least 3 months in the absence of disease progression or unacceptable toxicity. Patients may receive further treatment in the absence of disease progression.

Cohorts of 3-6 patients receive escalating doses of BMS-354825 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Once the MTD is determined, 20 additional patients receive treatment as in phase I at the MTD of BMS-354825.

Patients are followed for at least 30 days.

PROJECTED ACCRUAL: Approximately 50 patients (30 for phase I and 20 for phase II) will be accrued for this study within 12-18 months.

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnosis of Philadelphia chromosome positive, chronic phase chronic myelogenous leukemia (CML) meeting all of the following criteria*:
* Less than 15% blasts in peripheral blood and bone marrow
* Less than 20% basophils in peripheral blood
* Less than 30% blasts and promyelocytes in peripheral blood and bone marrow
* Platelet count at least 100,000/mm^3 NOTE: *Patients who previously met the criteria for accelerated phase or blast phase CML, responded to treatment, and currently meet the criteria for chronic phase CML are eligible
* Primary or acquired hematologic resistance to imatinib mesylate OR intolerance to imatinib mesylate defined as follows:
* Primary hematologic resistance is defined as failure to reach complete hematologic response (CHR) with a dose of 400 mg/day continued for at least 3 months

  * Patients with hematological progression (i.e., WBC at least 10,000/mm^3 and rising consistently on at least 2 consecutive measurements obtained at least 14 days apart) while receiving imatinib mesylate of 400 mg/day are eligible if they have received less than 3 months of therapy
* Acquired hematologic resistance is defined as achieving a CHR, but subsequently developing a rising WBC to at least 10,000/mm^3

  * WBC must be at least 10,000/mm^3 and rising on at least 2 measurements obtained at least 14 days apart with at least 1 of these measurements greater than 15,000/mm^3
* Intolerance is defined as having discontinued imatinib mesylate due to nonhematologic toxicity of any grade

  * CD4^+ T-cell count at least 350/mm^3
* 18 and over
* ECOG 0-1
* Life expectancy, At least 6 months.
* Hepatic

  * Bilirubin no greater than 1.5 mg/dL
  * ALT and AST no greater than 2.0 times upper limit of normal (ULN)
* Renal

  * Creatinine no greater than 1.5 times ULN
  * Potassium normal*
  * Magnesium normal*
  * Serum calcium or ionized calcium at least lower limit of normal NOTE: *Patients with low levels may be repleted to be eligible
* Negative pregnancy test
* Fertile patients must use effective contraception for 1 month before, during, and 1 month after study participation
* More than 14 days since prior interferon
* More than 14 days since prior cytarabine
* More than 3 days since prior hydroxyurea
* More than 28 days since other prior investigational or antineoplastic agents
* More than 7 days since prior imatinib mesylate
* At least 5 days or 5 half-lives since prior medications that inhibit platelet function, including the following:
* Aspirin
* Dipyridamole
* Epoprostenol
* Eptifibatide
* Clopidogrel
* Cilostazol
* Abciximab
* Ticlopidine
* At least 5 days or 5 half-lives since prior anticoagulants such as warfarin or heparin/low molecular weight heparin (e.g., danaparoid, dalteparin, tinzaparin, enoxaparin)
* At least 5 days or 5 half-lives since prior drugs accepted to have a risk of causing torsades de pointes, including the following:
* Class IA antiarrhythmic agents (e.g., quinidine, procainamide, or disopyramide)
* Class III antiarrhythmic agents (e.g., amiodarone, sotalol, ibutilide, or dofetilide)
* Macrolide antibiotics (e.g., erythromycin or clarithromycin)
* Antipsychotics (e.g., chlorpromazine, haloperidol, thioridazine, or pimozide)
* Tricyclic antidepressants
* Cisapride
* Bepridil
* Inapsine
* Methadone
* Arsenic
* Concurrent anagrelide for thrombocytosis due to CML allowed

Exclusion Criteria:

* extramedullary involvement (other than liver or spleen)
* significant bleeding disorder unrelated to CML
* acquired bleeding disorder within the past year (e.g., acquired antifactor VIII antibodies)
* congenital bleeding disorders (e.g., von Willebrand disease)
* uncontrolled or significant cardiovascular disease
* uncontrolled angina within the past 6 months
* congestive heart failure within the past 6 months
* myocardial infarction within the past 12 months
* history of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
* history of second or third degree heart block (may be eligible if patient has a pacemaker)
* diagnosed or suspected congenital long QT syndrome
* prolonged QTc interval on pre-entry EKG (i.e., greater than 450 msec)
* heart rate less than 50/minute on pre-entry EKG
* uncontrolled hypertension
* vasculitis
* pregnant or nursing
* gastrointestinal tract bleeding within the past 6 months
* connective tissue disorders
* other serious uncontrolled medical disorder or active infection that would impair the ability to receive study therapy
* dementia or altered mental status that would preclude giving informed consent
* evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, EKG, or clinical laboratory determinations unrelated to CML
* prisoners or patients who are compulsorily detained (e.g., involuntary incarceration for treatment of either a psychiatric or physical [e.g., infectious disease] illness)
* concurrent drugs accepted to have a risk of causing torsades de pointes
* other concurrent treatment for CML
* concurrent dolasetron or droperidol
* concurrent anticoagulants
* concurrent medications that inhibit platelet function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-11; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Sawyers, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Cortes J, Sawyers CL, Kantarjian HM, et al.: Long-term efficacy of dasatinib in chronic-phase CML: results from the phase I trial (CA180002). [Abstract] Blood 110 (11): A-1026, 2007.
- [Result] Talpaz M, Shah NP, Kantarjian H, Donato N, Nicoll J, Paquette R, Cortes J, O'Brien S, Nicaise C, Bleickardt E, Blackwood-Chirchir MA, Iyer V, Chen TT, Huang F, Decillis AP, Sawyers CL. Dasatinib in imatinib-resistant Philadelphia chromosome-positive leukemias. N Engl J Med. 2006 Jun 15;354(24):2531-41. doi: 10.1056/NEJMoa055229. PMID 16775234
- [Result] Talpaz M, Kantarjian HM, Paquette R, et al.: A phase I study of BMS-354825 in patients with imatinib-resistant and intolerant chronic phase chronic myeloid leukemia (CML): results from CA180002. [Abstract] J Clin Oncol 23 (Suppl 16): A-6519, 564s, 2005.